CLINICAL TRIAL: NCT03909958
Title: The Impact of Electroacupuncture on Clinical Effect,Brain Structural and Functional Changes in Patients With Spinal Cord Injury:A Randomized Controlled Study Based on Multi-mode MRI
Brief Title: The Impact of Electroacupuncture on Clinical Effect,Brain Structural and Functional Changes on Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Ruijie Ma, Professor,Vice president of the Third Affiliated hospital of Zhejiang Chinese Medical University, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019ZZ013; NCT03909087 (obsolete NCT alias)
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injury; electroacupuncture; Brain Structure and Function; Multi-mode Magnetic Resonance Imaging
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture+Routine rehabilitation training Group (Other): 42 patients will receive both electroacupuncture（HANS100A）therapy and routine rehabilitation training.
  Interventions: Other: Electroacupuncture+Routine rehabilitation training Group
- Routine rehabilitation training Group (Other): 42 patients will receive simple routine rehabilitation training.
  Interventions: Behavioral: Routine rehabilitation training Group

INTERVENTIONS:
Other: Electroacupuncture+Routine rehabilitation training Group — Electroacupuncture： Major acupoints: Jiaji points. With urinary and stool dysfunction:+Shenshu (BL23) ,Huiyang(BL35).
  Localization:Jiaji points of the upper 1 and the lower 1 segment of the Spinal cord injury plane, a total of 4 points.
  Operation: Insert Jiaji points By using Hwato-brand disposable acupuncture needles(0.30mm*50mm), with 0.5 inch from the median line and a depth of 50 to 60mm with perpendicular insertion.Then, participants will receive electroacupuncture treatment by connecting Han's pain irritant instrument (HANS100A) for 30min with the stimulation frequency of 2 /100 Hz and intensity of 1-2mA. Once a day, 5 days a week and rest 2 days, a week is one course and the duration need 12 courses.
  Routine rehabilitation training:
  Same as Routine rehabilitation training Group.
  Arms: Electroacupuncture+Routine rehabilitation training Group
Behavioral: Routine rehabilitation training Group — Routine rehabilitation training:
  Participants with good spinal stability will receive sitting training as early as possible, and will carry out standing training if participants had no adverse reactions (postural hypotension, etc.) after sitting training. Muscle strength training will be performed in recovery phase, and functional movement training will be selected according to participants' conditions. Functional movement training and transfer training will be performed for 20min each time and once a day;Standing and walking training, 2 times a day, 30min each time.
  Arms: Routine rehabilitation training Group

SUMMARY:
Spinal cord injury (SCI) is a kind of severe disease with high morbidity and complications. At present, electroacupuncture has certain advantages in treating motor sensory dysfunction, neuropathologic pain, neurogenic bladder and intestinal dysfunction after spinal cord injury. However, previous clinical studies of acupuncture neglected the brain, which is closely related to the structure and function of spinal cord.So,the aim of this study is to observe and analyse the impact of the changes of gray and white matter volume on whole brain and brain functional re-establish,to reveal the neuroimaging mechanism of improving the motor sensory functions of patients with spinal cord injury, and to provide a theoretical basis for the clinical application of electroacupuncture.

ELIGIBILITY:
1.Aged 18-75 years no matter the gender 2.14 days to 3 months after the onset of SCI 3.Patients with cervical, thoracic or lumbar spinal cord injuries 4.SCI classified as B, C, or D grade on the ASIA impairment scale(AIS), that is incomplete SCI (iSCI) 5.Patients with grade 1-3 muscle strength of lower limbs 6.Right-handed 7.Patients who submitted written informed consent

Exclusion Criteria:

1. Contraindication to MRI scanning such as metal in the body, pacemaker
2. Severe structural asymmetry or lesions in the brain
3. Complications that may affect neurologic examination, such as severe peripheral nerve injury, limb fractures, and heterotopic ossification around the joints
4. With complex injury such as traumatic brain injury, organ injury, unstable vital signs or disturbance of consciousness
5. With severe primary diseases such as heart, liver, kidney and hematopoietic system
6. Patients with SCI due to myelitis, multiple sclerosis, vascular malformation caused spinal cord hemorrhage, intraspinal tumors, etc.
7. Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2019-11-26 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Brain structure data(Changes of gray and white matter volume on whole brain based on fMRI) | Before intervention; the end of the 3rd month when treatment finished.
  The 3D MPRAGE image data collected by fMRI will be recorded and exported on a CD, and then will be processed and analyzed by VBM8.
Brain function data(Changes of ALFF value and FC value of the whole brain based on fMRI) | Before intervention; the end of the 3rd month when treatment finished.
  The REST fMRI image data will be recorded and exported to a CD, and then will be processed and analyzed with REST software and seed point method to calculate the ALFF value and FC value of the whole brain.

SECONDARY OUTCOMES:
Change in ASIA (American Spinal Injury Association) grade | Before intervention; after 6 weeks of treatment;the end of the 3rd month when treatment finished;fellow-up period at the 6th month.
  To assess the motor function and the sensory function. The motor function will be evaluated according to the scores of five key muscles and muscle strength in both lower limbs.This score can reflect the degree of neurological impairment associated with the SCI, with lower score indicating greater impairment. Score ranges from 0-25 for each extremity, with maximum scores of 50 for the upper limbs and 50 for the lower limbs.
  The sensory function will be evaluated according to the scores of bilateral pain sensation and tactile sensation in 14 key sensory points in both lower limbs. This score can reflect the degree of neurological impairment associated with the SCI, with lower score indicating greater impairment. Score ranges from 0-56 points each for light touch and pin prick (sharp/dull discrimination) modalities, with a maximum total score of 112 points per side of the body.
Change in Modified Ashworth Scale(MAS) | Before intervention; after 6 weeks of treatment;the end of the 3rd month when treatment finished;fellow-up period at the 6th month.
  To assess the muscle tone.MAS grades as follows:
  0: No increase in muscle tone.1: Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is(are) moved in flexion or extension.1+: Slight increase in muscle tone, manifested by a catch followed by minimal resistance through the remainder of the range of motion but the affected part(s) is(are) easily moved.2: More marked increase in muscle tone through most of the range of movement, but the affected part(s) is easily moved.3: Considerable increases in muscle tone, passive movement difficult.4: Affected part(s) is (are) rigid in flexion or extension.
Change in Modified Barthel Index(MBI) | Before intervention; after 6 weeks of treatment;the end of the 3rd month when treatment finished;fellow-up period at the 6th month.
  To assess the ability of the patient to perform daily activities.It comprises 10 items regarding activities of daily living and mobility and assesses feeding, transfer from wheelchair to bed and back, self-care, bathing, walking, climbing stairs, dressing, and bladder and bowel continence. Scoring is based on whether the patient requires help or not in performing any of the above mentioned activities.Scale range: 0-100.Higher score means better function and less dependence.

CONTACTS AND LOCATIONS:
Overall Officials: Ruijie Ma, Dr., Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (1):
- The Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hunter Revell SM. Symptom clusters in traumatic spinal cord injury: an exploratory literature review. J Neurosci Nurs. 2011 Apr;43(2):85-93. doi: 10.1097/jnn.0b013e31820c2533. PMID 21488582
- [Background] National Spinal Cord Injury Statistical Center. Spinal cord injury facts and figures at a glance. J Spinal Cord Med. 2013 Jan;36(1):1-2. doi: 10.1179/1079026813Z.000000000136. No abstract available. PMID 23433327
- [Background] Heo I, Shin BC, Kim YD, Hwang EH, Han CW, Heo KH. Acupuncture for spinal cord injury and its complications: a systematic review and meta-analysis of randomized controlled trials. Evid Based Complement Alternat Med. 2013;2013:364216. doi: 10.1155/2013/364216. Epub 2013 Feb 17. PMID 23476688
- [Background] Rekand T, Hagen EM, Gronning M. Chronic pain following spinal cord injury. Tidsskr Nor Laegeforen. 2012 Apr 30;132(8):974-9. doi: 10.4045/tidsskr.11.0794. English, Norwegian. PMID 22562333
- [Background] Shin BC, Lee MS, Kong JC, Jang I, Park JJ. Acupuncture for spinal cord injury survivors in Chinese literature: a systematic review. Complement Ther Med. 2009 Oct-Dec;17(5-6):316-27. doi: 10.1016/j.ctim.2009.09.001. Epub 2009 Oct 21. PMID 19942112
- [Background] Buss A, Brook GA, Kakulas B, Martin D, Franzen R, Schoenen J, Noth J, Schmitt AB. Gradual loss of myelin and formation of an astrocytic scar during Wallerian degeneration in the human spinal cord. Brain. 2004 Jan;127(Pt 1):34-44. doi: 10.1093/brain/awh001. Epub 2003 Oct 8. PMID 14534158
- [Background] Hains BC, Black JA, Waxman SG. Primary cortical motor neurons undergo apoptosis after axotomizing spinal cord injury. J Comp Neurol. 2003 Jun 9;462(3):328-41. doi: 10.1002/cne.10733. PMID 12794736
- [Background] Kim BG, Dai HN, McAtee M, Vicini S, Bregman BS. Remodeling of synaptic structures in the motor cortex following spinal cord injury. Exp Neurol. 2006 Apr;198(2):401-15. doi: 10.1016/j.expneurol.2005.12.010. Epub 2006 Jan 26. PMID 16443221
- [Background] Wu J, Zhao Z, Sabirzhanov B, Stoica BA, Kumar A, Luo T, Skovira J, Faden AI. Spinal cord injury causes brain inflammation associated with cognitive and affective changes: role of cell cycle pathways. J Neurosci. 2014 Aug 13;34(33):10989-1006. doi: 10.1523/JNEUROSCI.5110-13.2014. PMID 25122899
- [Background] Altamura AC, Maggioni E, Dhanoa T, Ciappolino V, Paoli RA, Cremaschi L, Prunas C, Orsenigo G, Caletti E, Cinnante CM, Triulzi FM, Dell'Osso B, Yatham L, Brambilla P. The impact of psychosis on brain anatomy in bipolar disorder: A structural MRI study. J Affect Disord. 2018 Jun;233:100-109. doi: 10.1016/j.jad.2017.11.092. Epub 2017 Nov 29. PMID 29223329
- [Background] Saricicek A, Yalin N, Hidiroglu C, Cavusoglu B, Tas C, Ceylan D, Zorlu N, Ada E, Tunca Z, Ozerdem A. Neuroanatomical correlates of genetic risk for bipolar disorder: A voxel-based morphometry study in bipolar type I patients and healthy first degree relatives. J Affect Disord. 2015 Nov 1;186:110-8. doi: 10.1016/j.jad.2015.06.055. Epub 2015 Jul 26. PMID 26233321
- [Background] Hutton C, De Vita E, Ashburner J, Deichmann R, Turner R. Voxel-based cortical thickness measurements in MRI. Neuroimage. 2008 May 1;40(4):1701-10. doi: 10.1016/j.neuroimage.2008.01.027. Epub 2008 Feb 1. PMID 18325790
- [Background] Benetti S, Pettersson-Yeo W, Hutton C, Catani M, Williams SC, Allen P, Kambeitz-Ilankovic LM, McGuire P, Mechelli A. Elucidating neuroanatomical alterations in the at risk mental state and first episode psychosis: a combined voxel-based morphometry and voxel-based cortical thickness study. Schizophr Res. 2013 Nov;150(2-3):505-11. doi: 10.1016/j.schres.2013.08.030. Epub 2013 Sep 29. PMID 24084578
- [Background] Freund P, Weiskopf N, Ward NS, Hutton C, Gall A, Ciccarelli O, Craggs M, Friston K, Thompson AJ. Disability, atrophy and cortical reorganization following spinal cord injury. Brain. 2011 Jun;134(Pt 6):1610-22. doi: 10.1093/brain/awr093. Epub 2011 May 17. PMID 21586596
- [Background] Jurkiewicz MT, Crawley AP, Verrier MC, Fehlings MG, Mikulis DJ. Somatosensory cortical atrophy after spinal cord injury: a voxel-based morphometry study. Neurology. 2006 Mar 14;66(5):762-4. doi: 10.1212/01.wnl.0000201276.28141.40. PMID 16534122
- [Background] Ma R, Liu X, Clark J, Williams GM, Doi SA. The Impact of Acupuncture on Neurological Recovery in Spinal Cord Injury: A Systematic Review and Meta-Analysis. J Neurotrauma. 2015 Dec 15;32(24):1943-57. doi: 10.1089/neu.2014.3866. Epub 2015 Aug 28. PMID 26079978